CLINICAL TRIAL: NCT05077384
Title: An Open-Label Study of Surufatinib in Japanese Patients With Neuroendocrine Tumors
Brief Title: Open-label Study of Surufatinib in Japanese Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-012-00JP1
Expanded Access: NCT04814732 (No longer available)
Record Dates: First submitted 2021-09-20; First posted 2021-10-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Tumors; Non-hematologic Malignancy
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Surufatinib (Experimental): Oral surufatinib 300 mg once daily in treatment cycles of 28 days starting at Cycle 1 Day1
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300 mg oral once daily
  Other Names: HMPL-012; sulfatinib

SUMMARY:
This is a phase 1/2, open-label, multi-centre study of surufatinib in patients with unresectable, locally advanced, or recurrent nonhematologic malignancies who do not respond or are intolerant to standard of care.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the tolerability and efficacy of surufatinib in Japanese patients.

The study will be conducted in 2 parts:

* Part 1 - evaluation of tolerability and safety of surufatinib and confirmation of the recommended clinical dose in Japanese patients with nonhematologic malignancies
* Part 2 - evaluation of antitumor activity and confirmation of tolerability of surufatinib in Japanese patients with NETs

All patients will be treated with oral surufatinib 300 mg QD in treatment cycles of 28 days starting on Cycle 1 Day 1.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically documented disease as follows:

   1. Part 1: unresectable, locally advanced or metastatic nonhematologic malignancy that is relapsed/refractory to or intolerant of established therapies known to provide clinical benefit
   2. Part 2: locally advanced or metastatic, low (grade 1) or intermediate (grade 2) grade NETs that have been previously treated with at least 1 line of systemic therapy
2. Has radiologic evidence of progressive tumour within 12 months of study enrolment
3. Is willing and able to provide informed consent
4. Is ≥20 years of age
5. Has measurable lesions according to RECIST Version 1.1
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Female patients of childbearing potential and male patients with partners of childbearing potential agree to use a highly effective form(s) of contraception

Key Exclusion Criteria:

1. Women who are pregnant and lactating, or possibly pregnant.
2. Has a history of interstitial lung disease (ILD)/noninfectious pneumonitis, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
3. Known active viral hepatits
4. Has an AE due to previous anti-tumour therapy that has not recovered to ≤CTCAE Grade 1, except alopecia and peripheral neurotoxicity with ≤CTCAE Grade 2 caused by platinum chemotherapy
5. Uncontrollable hypertension, defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, despite antihypertensive medication
6. Gastrointestinal disease or condition within 6 months prior to first dose
7. Has a history or presence of a serious haemorrhage (>30 mL within 3 months) or haemoptysis (>5 mL blood within 4 weeks)
8. Clinically significant cardiovascular disease.
9. Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of stable disease (SD) for 14 days or longer; patients requiring steroids within 4 weeks prior to start of study treatment will be excluded.
10. A high risk of bleeding at screening due to tumour invasion into major vessels, such as pulmonary artery, the superior vena cava, or the inferior vena cava, as determined by investigators.
11. Has arterial thrombosis or deep venous thrombosis within 6 months prior to first dosing, or thromboembolic events (including stroke and/or transient ischaemic attack) within 12 months prior to first dosing.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of treatment-emergent adverse events (TEAEs) graded by the Investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0). | Up to 2 years
  To evaluate surufatinib-related adverse events in patients with NETs
Part 2: Objective response rate. This will be assessed on the proportion of participants with partial response or complete response as determined by the Investigator based on RECIST v1.1 | Up to 2 years
  The primary outcome of part 2 will be objective response rate in patients with NETs when treated with surufatinib

SECONDARY OUTCOMES:
Observed plasma concentrations of surufatinib which will be assessed by the Cmax, tmax, AUC, Cmin and CL/F | Up to 2 years
  Blood sampling will be taken to measure levels of the study drug
Progression Free Survival (PFS) which is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator based on RECIST v1.1, or death from any cause, whichever occurs first | Up to 2 years
  The duration between the enrollment date and the first disease progression (PD) or death (whichever comes first).
Duration of Response (DOR) which will be defined as the time from the first response to disease progression documented after treatment initiation or death, whichever occurs first. DOR will include CR, CR plus CRi, overall response (OR), and CR plus CRh. | Up to 2 years
  The duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, MD, Study Director — Hutchmed
Locations (12):
- Japan (12):
  - Kyushu University Hospital, Fukuoka
  - Fukuoka Sanno Hospital, Fukuoka
  - Kagawa University Hospital, Kagawa
  - National Cancer Centre Hospital East, Kashiwa-shi
  - Kyoto University Hospital, Kyoto
  - Kyorin University Hospital, Mitaka
  - Aichi Cancer Centre, Nagoya
  - Kansia Electric Power Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - National Cancer Centre Hospital, Tokyo
  - Yokohama City University Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: No